CLINICAL TRIAL: NCT05985694
Title: A Single-blind (Patient-blind), Randomized, Placebo-controlled, Intranasal Administration Study on Mechanisms and Potential Efficacy of AD17002 in Subjects With Poorly Controlled, Moderate to Severe Eosinophilic Asthma
Brief Title: AD17002 Treating Poorly Controlled, Moderate to Severe Eosinophilic Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advagene Biopharma Co. Ltd. (Industry)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADV_Asthma_17002-1
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Eosinophilic Asthma
Keywords: LTh(αK), Type I/III Interferon, Immunomodulator, epithelial
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — heat-labile enterotoxin, E coli

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 Placebo (Placebo Comparator): Formulation buffer
  Interventions: Drug: Placebo
- Cohort 1 Low dose (Experimental): Formulation buffer + 10 μg AD17002
  Interventions: Drug: AD17002
- Cohort 2 Placebo (Placebo Comparator): Formulation buffer
  Interventions: Drug: Placebo
- Cohort 2 High dose (Experimental): Formulation buffer + 20 μg AD17002
  Interventions: Drug: AD17002

INTERVENTIONS:
Drug: AD17002 — The dosing days of AD17002 are: Days 1, 4, 8, 11, 15, 18, 22, 25, 29, and 32.
  Other Names: LTh(αK)
  Arms: Cohort 1 Low dose; Cohort 2 High dose
Drug: Placebo — Formulation buffer. Dosing days: 1, 4, 8, 11, 15, 18, 22, 25, 29, 32.
  Other Names: Formulation buffer
  Arms: Cohort 1 Placebo; Cohort 2 Placebo

SUMMARY:
This clinical trial aims to investigate patients with poorly controlled, moderate to severe eosinophilic asthma. The main questions it seeks to answer are

1. Could the AD17002 intranasal immunomodulator improve the clinical condition of eosinophilic asthmatic patients?
2. Could patients self-administer AD17002 via the intranasal route?
3. Is the AD17002 at multiple doses safe for asthmatic patients?
4. Participants will be asked to self-administer two doses per week for a total of 6 weeks (11 doses). A diary on AD17002 usage, adverse events, and reliever medication will be recorded.

DETAILED DESCRIPTION:
This study was conducted to determine the potential efficacy and mechanism of AD17002 as an immunomodulator in attenuating the severity of clinical manifestations in patients with unstable, moderate-to-severe eosinophilic asthma. Patients with clinical history and ongoing eosinophilic asthma will be randomly assigned to either AD17002 (10 μg or 20 μg) or placebo, per 3-4 days, in a 1:1 ratio, in a single-blinded (patient-blinded) fashion. The nasal administration will be self-administered by participants. Progression and improvement in asthmatic symptoms will be recorded. All study subjects will sign ethics committee-approved informed consent forms before participating in any trial-related activities. Subjects who participate in this trial of AD17002 will provide information about the dosing, efficacy, and safety of the new indication that will guide its future clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Subject 20-80 years of age on the day of signing informed consent
2. Subject who is not a current smoker with poorly controlled, moderate to severe eosinophilic asthma based on GINA 2022 criteria.
3. The subject is diagnosed with asthma.
4. Subjects who have the post-bronchodilator reversibility of Forced expiratory volume 1 (FEV1) of ≥ 12% and ≥ 200 mL in response to a SABA at the screening visit or documented in the medical chart within 3 months of the screening visit.
5. Subjects who have ≥3% eosinophil counts in the induced sputum within 7 days of Visit 1.
6. Subjects with ACT scores ≤ 19 under regular low to moderate-dose inhaled corticosteroids (ICS) and/or a combination with inhaled long-acting beta 2 agonists for at least 3 months before the Screening Visit.
7. Have a negative serum pregnancy test at the screening, and randomization visits (female subjects of childbearing potential). A female subject who is of reproductive potential agrees to remain abstinent or use (or have their partner use) an acceptable method of birth control within the projected duration of the trial. Acceptable birth control methods are intrauterine devices, hormonal contraception, diaphragm with spermicide, contraceptive sponge, condoms, and vasectomy, as per local regulations or guidelines.
8. A female subject who is not of reproductive potential is eligible without requiring the use of contraception. A female subject who is not of reproductive potential is defined as one who has either
9. Reached natural menopause (defined as 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone levels in the postmenopausal range as determined by the laboratory, or 12 months of spontaneous amenorrhea),
10. Six weeks postsurgical documented total hysterectomy and/or bilateral salpingo-oophorectomy, or
11. Bilateral tubal ligation.
12. Subject or the subject's legal representative understands the trial procedures, alternative treatments available, and risks involved with the trial, and voluntarily agrees to participate by giving written informed consent.
13. Provide written informed consent for the trial and be willing to adhere to dose and visit schedules.

Exclusion Criteria:

1. Subjects with serious underlying chronic illness or severe systemic disease, including SLE, malignant diseases, uremia and heart failure, or abnormal liver function.
2. Subjects without a recent respiratory tract infection within 3 weeks before the study.
3. Subjects without a recent COVID-19 infection within 1 month before study.
4. Subjects with clinically important lung disease, including but not limited to COPD (Chronic Obstructive Pulmonary Disease), chronic respiratory infection, lung cancer, etc.
5. Arrhythmia, myocardial infarction, or stroke in the last 3 months.
6. Active COVID-19 disease (SARS-CoV-2 Lateral flow tests (LFA)-positive) at Screening.
7. A clinical history of persistent allergic asthma or rhinitis caused by an allergen to which the subject is regularly exposed and sensitized.
8. A clinical history of active chronic sinusitis (> 3 months).
9. Any clinically relevant chronic disease (>=3 months duration) (e.g. cystic fibrosis, malignancy, renal or hepatic insufficiency).
10. Subject with a documented history of Bell's palsy.
11. The subject has any nasal condition that could confound the efficacy or safety assessments.
12. Immunosuppressive treatment (ATC code L04 or L01) within 3 months before the screening visit (except the specified concomitant medications for allergy and asthma symptoms).
13. Has unstable or severe asthma, as judged by the clinical Investigator, or a subject who has experienced a life-threatening asthma attack or an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids (but allowing SABA) at any time within the last 3 months before Screening Visit.
14. Has asthma requiring high-dose oral corticosteroid (OCS) within the last 3 months before Screening Visit.
15. Has a history of anaphylaxis with cardiorespiratory symptoms with prior immunotherapy, unknown cause, or inhalant allergen.
16. Is pregnant or expecting to conceive within the projected duration of the trial.
17. Is nursing at randomization and within the projected duration of the trial?
18. Has had previous exposure to the study drug or Flu Vaccine AD07030.
19. The subject is receiving ongoing treatment with any specific immunotherapy at the time of the Screening Visit.
20. Has a known history of allergy, hypersensitivity, or intolerance to investigational medicinal products, rescue medications, or self-injectable epinephrine.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
FEV1 improvement | Day 1 to Day 78
  Lung function tests with spirometry

SECONDARY OUTCOMES:
Change to the use of Short-Acting Beta Agonists (SABA) | Day 1 to Day 78
  The number of use of rescue Short-Acting Beta Agonists
Fractional exhaled nitric oxide (FeNO) change | Day 1 to Day 78
  Change to the FeNO levels
changes of sputum eosinophil counts | Day 1 to Day 78
  Change to the induced sputum eosinophils' count
Asthma Control Test (ACT) scores improvement | Day 1 to Day 78
  Change to the ACT scores. A maximum score of 25 points indicates complete asthma control. A score between 20 and 25 represents well controlled asthma, while a score of 19 or below represents not well controlled asthma, and a score less than 16 indicates very poorly controlled asthma.
Corticosteroid used to control asthma | Day 1 to Day 78
  Numbers of corticosteroid used, inhaled or oral
Immunological biomarkers of sputum | Day 1 to Day 78
  Changes in the concentration of sputum IL-4, -5, -13, IFN-α, eosinophil peroxidase (EPO), eosinophil cationic protein (ECP) from the baseline
Immunological biomarkers of serum | Day 1 to Day 78
  Change of concentration from baseline of induced serum IL-4, -5, -13
Peripheral eosinophil count | Day 1 to Day 78
  Change of cell numbers from baseline of peripheral eosinophil count
Adverse events_clinical visit | Day 1 to Day 36 and Day 78
  Clinical visit and check up by physicians
Adverse events-Diary | Day 1 to Day 78
  Patient self report adverse events via diary

CONTACTS AND LOCATIONS:
Overall Officials: Yushen Hsu, Ph.D., Study Chair — Advagene Biopharma; Han-Pin Kuo, MD. Ph.D., Study Director — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan